CLINICAL TRIAL: NCT06062628
Title: Neurophysiological Effect of Ketamine in Patients With Severe Traumatic Brain Injury
Brief Title: Ketamine in Severe Traumatic Brain Injury
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anna Bashmakov, Neurology - Neuro Critical Care Fellow, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0805
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; Traumatic Encephalopathy
Keywords: ketamine; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine Intervention Arm (Experimental): A single dose of 0.5 mg/kg (actual body weight) of ketamine will be administered intravenously. Ketamine will be administered in addition to the patient's existing analgesia, sedation and other medicines as a part of their routine treatment.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Administration of ketamine with subsequent measurement of intracranial pressure and brain tissue oxygenation

SUMMARY:
Traumatic brain injury (TBI) accounts for approximately 2.5 million visits to emergency departments in the United States each year. After decades of research, management strategies for severe TBI (sTBI) patients are still evolving. Optimizing intracranial pressure (ICP) and cerebral perfusion pressure (CPP) are paramount in the management of these patients and placement of these monitors is the current standard-of-care. However, monitoring brain oxygenation (PbtO2) with invasive intraparenchymal monitors is currently under investigation in the management of severe TBI and placement of these monitors is gaining widespread use. This has opened the door for the use of tiered therapy to optimize ICP and PbtO2 simultaneously. Current evidence indicates that correction of ICP, CPP and PbtO2 in sTBI requires optimized analgesia and sedation. Ketamine is one of the few drugs available that has both sedative and analgesic properties and does not commonly compromise respiratory drive like opioids and sedative-hypnotics. However, traditionally, ketamine has been viewed as contraindicated in the setting of TBI due to concerns for elevation in ICP. Yet, new data has cast this long-held assumption into significant doubt. Hence the present pilot study will characterize the neurophysiological response to a single dose of ketamine in critically-ill TBI patient with ICP and PbtO2 monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Severe traumatic brain injury
* Placement of intracranial monitor for measurement of intracranial pressure and brain tissue oxygenation
* Age greater than or equal to 18 years

Exclusion Criteria:

* Documented allergy to ketamine
* Sinus tachycardia with sustained heart rate >120
* Any episode of non-sinus tachycardia
* Documented history of schizophrenia
* Systolic blood pressure > 180, diastolic blood pressure > 120
* Documented episode(s) of ICP elevations >25 mm Hg sustained greater than 5 minutes within 24 hours
* Similar episodes as above of PbtO2 <15 mmHg
* Positive pregnancy test and/or is currently breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intracranial Pressure (ICP, measured by external ventricular drain and/or ICP monitor) | 3 hours
  Measurement of pressure within the rigid skill, with values greater than 22 mm Hg sustained proven to be injurious in patients with traumatic brain injury
Brain tissue oxygenation (measured by intracranial oxygen probe) | 3 hours
  Measurement of the concentration of oxygen within the brain tissue, with values less than 20 mmHg sustained proven to be injurious in patients with traumatic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bashmakov, D.O., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No